CLINICAL TRIAL: NCT05457673
Title: Subcostal Temporary Extravascular Pacing IV (STEP IV) Study
Acronym: STEP IV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AtaCor Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: DOC-10200
Record Dates: First submitted 2022-07-06; First posted 2022-07-14 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Conduction Defect
Keywords: Temporary Ventricular Pacing; Extravascular
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AtaCor EV Temporary Pacing Lead System (Experimental): Subjects implanted with the AtaCor StealthTrac Lead Model AC-1013
  Interventions: Device: AtaCor StealthTrac Lead

INTERVENTIONS:
Device: AtaCor StealthTrac Lead — Subjects will receive the AtaCor StealthTrac Lead being evaluated in the study.

SUMMARY:
The STEP IV Study is a prospective, single-center, non-randomized, single-arm study without concurrent or historical controls. The objective of the study is to generate safety and performance data of the latest AtaCor EV Temporary Pacing Lead System to support the development of a future pivotal study with an indication limited to a maximum of 7 days.

DETAILED DESCRIPTION:
The primary safety objective is freedom from Adverse Device Effects (ADE). The primary performance objective is summary statistics for pacing capture threshold, impedance, and sensed R-wave amplitude with the StealthTrac Lead from insertion through removal.

One (1) Investigational Site in Paraguay will participate with up to 16 subjects enrolled in the study. Subjects indicated for a closed-chest cardiac invasive procedure will be eligible for participation. Subjects undergoing a qualifying index procedure will have a Model AC-1013 StealthTrac Lead inserted and evaluated over the follow-up period (up to 7 days post procedure). Study participation requires 2 to 7 days with the Study Lead inserted. Following Study Lead removal, a final follow-up will be performed 27-33 days after lead insertion to assess for any latent Adverse Events. Subjects remain enrolled until completion of the 30-Day Follow Up.

The maximum duration for study participation is 33 days. The Study is expected to last up to 3 months after first enrollment: Enrollment and follow-up (1 month) and final report (2 months).

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years old
2. Indicated for closed-chest cardiac invasive procedure (e.g., transcatheter valve replacement, balloon valvuloplasty, permanent pacemaker implantation and pacing lead extractions/revisions)

Exclusion Criteria:

1. BMI ≥ 35 kg/m2
2. Septic shock
3. Severe anemia
4. Acute coronary syndrome within past 90 days
5. NYHA IV Functional Classification of heart failure within past 90 days
6. Circumstances that prevent data collection or follow-up (e.g., inability to perform a short walk with the Holter monitor)
7. Participation in any concurrent clinical study without prior written approval from the Sponsor
8. Inability or unwillingness to provide informed consent to participate in the Study

   Known prior history for any of the following:
9. Median or partial sternotomy
10. Surgery with disruption of the lung, pericardium or connective tissue between the sternum and pericardium
11. Significant anatomic derangement of or within the thorax (e.g., pectus excavatum, significant scoliosis)
12. Thoracic radiation therapy, pneumothorax, pneumomediastinum or other medical treatments/conditions which may complicate the AtaCor EV Temporary Pacing Lead System insertion procedure
13. Pericardial disease, pericarditis and mediastinitis
14. Medical treatments, surgeries or conditions that increase the potential for pericardial adhesions
15. FEV1 < 1 liter
16. Surgically corrected congenital heart disease (not including catheter-based procedures)
17. Allergies to the device materials such as stainless steel, titanium, platinum, iridium, polyethylene, polyurethane, polycarbonate, and silicone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-08-17 (Actual); Primary Completion 2022-09-22 (Actual); Study Completion 2022-10-20 (Actual)

PRIMARY OUTCOMES:
Freedom from ADEs | Up to 7 days post-implant
  Freedom from Adverse Device Effects (ADEs)
Pacing Capture Threshold (V or mA) | Up to 7 days post-implant
  Summary statistics for pacing capture threshold with the StealthTrac Lead from insertion through removal
Impedance (Ohms) | Up to 7 days post-implant
  Summary statistics for impedance with the StealthTrac Lead from insertion through removal
Sensed R-Wave Amplitude (mV) | Up to 7 days post-implant
  Summary statistics for sensed R-wave amplitude with the StealthTrac Lead from insertion through removal

CONTACTS AND LOCATIONS:
Overall Officials: Martin C Burke, DO, Principal Investigator — AtaCor Medical, Inc.
Locations (1):
- Sanatorio Italiano, Asunción, Paraguay

IPD SHARING:
Plan to Share IPD: No